CLINICAL TRIAL: NCT00630279
Title: A Multi-center, Single-blind, Parallel-design, Randomized, Placebo-controlled, Dose-ranging Study to Evaluate Oral Recombinant Microbial Lipase Efficacy in Patients With Pancreatic Exocrine Insufficiency Due to Chronic Pancreatitis
Brief Title: Dose-ranging Study to Evaluate Efficacy of SLV339 in Pancreatic Exocrine Insufficiency Due to Chronic Pancreatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This trial discontinued March 7,2009 due to high screen failure rate.
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Veronika von Hahn, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S339.2.001; 2007-000375-42
Record Dates: First submitted 2008-02-22; First posted 2008-03-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Pancreatic Exocrine Insufficiency Due to Chronic Pancreatitis
Keywords: pancreatic exocrine insufficiency; chronic pancreatitis
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Pancreatitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: Recombinant Microbial Lipase SLV339
- 3 (Experimental)
  Interventions: Drug: Recombinant Microbial Lipase SLV339
- 4 (Experimental)
  Interventions: Drug: Recombinant Microbial Lipase SLV339

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: 1
Drug: Recombinant Microbial Lipase SLV339 — oral, 150 mg/d, 7 days treatment
  Arms: 2
Drug: Recombinant Microbial Lipase SLV339 — oral, 300 mg/d, 7 days treatment
  Arms: 3
Drug: Recombinant Microbial Lipase SLV339 — oral, 600 mg/d, 7 days treatment
  Arms: 4

SUMMARY:
This study is to estimate the efficacy of a number of doses in patients with pancreatic insufficiency

ELIGIBILITY:
Inclusion Criteria:

* Subject > 18 years;
* Pancreatic exocrine insufficiency confirmed and documented in medical history by either a pathophysiological direct or indirect pancreatic function test or clinical symptoms of steatorrhea stool fat that resolved or improved substantially upon pancreatic enzyme supplementation;
* Patients on a stable daily dose of pancreatic enzymes for 3 months;
* Subjects with CP with or without partial pancreatectomy due to CP, confirmed in medical history by either CT , ERCP, plain film with pancreatic calcifications, ultra-sonography (calcifications, duct dilatation), magnetic resonance pancreatography, endoscope ultrasound, other radiological diagnosis captured by tools such as Cambridge classification and /or histology;
* CFA < 80% at time of randomization

Exclusion Criteria:

* Evidence of major surgery (except gall bladder removal or appendectomy) or other relevant diseases as revealed by history, physical examination, and laboratory assessments which may interfere with the absorption, distribution, metabolism or elimination of the study drug or constitute a risk factor when taking the study medication;
* Investigational drug intake within 90 days prior to the pre-assessment visit;
* Ileus or acute abdomen;
* Allergic disease such as hypersensitivity pneumonitis, aspergillus mediated asthma or allergic broncho-pulmonary aspergillosis;
* Stenosis or regurgitation of the esophagus or stomach;
* Known HIV infection, acute phase of CP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
CFA (Coefficient of Fat Absorption) | from baseline to end of 7 days treatment

SECONDARY OUTCOMES:
CNA, stool fat, stool weight, nutritional parameters, clinical symptomatology | from baseline to end of 7 days treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (50):
- Czechia (6):
  - Site 4206, Brno
  - Site 4203, Hradec Králové
  - Site 4202, Prague
  - Site 4205, Prague
  - Site 4201, Tábor
  - Site 4204, Ústí nad Orlicí
- Denmark (3):
  - Site 4503, Herning
  - Site 4502, Hvidovre
  - Site 4501, Odense
- Hungary (15):
  - Site 3612, Békéscsaba
  - Site 3607, Budapest
  - Site 3614, Budapest
  - Site 3615, Debrecen
  - Site 3602, Dunaújváros
  - Site 3610, Eger
  - Site 3604, Gyula
  - Site 3606, Pécs
  - Site 3613, Sopron
  - Site 3609, Szeged
  - Site 3601, Szekszárd
  - Site 3611, Szentes
  - Site 3608, Tatabánya
  - Site 3603, Vác
  - Site 3605, Zalaegerszeg
- Latvia (5):
  - Site 3702, Daugavpils
  - Site 3701, Riga
  - Site 3703, Riga
  - Site 3704, Riga
  - Site 3705, Riga
- Poland (13):
  - Site 4808, Bialystok
  - Site 4809, Gdansk
  - Site 4810, Gdansk
  - Site 4805, Katowice
  - Site 4811, Lodz
  - Site 4807, Poznan
  - Site 4814, Poznan
  - Site 4802, Skierniewice
  - Site 4804, Sopot
  - Site 4801, Warsaw
  - Site 4806, Warsaw
  - Site 4812, Wroclaw
  - Site 4813, Wroclaw
- Russia (5):
  - Site 0901, Moscow
  - Site 0904, Moscow
  - Site 0908, Moscow
  - Site 0909, Moscow
  - Site 0910, Moscow
- Sweden (3):
  - Site 4602, Gothenburg
  - Site 4603, Stockholm
  - Site 4601, Umeå